CLINICAL TRIAL: NCT00278148
Title: A Phase I/II Trial of Neoadjuvant Paclitaxel, Carboplatin and OSI-774 (Tarceva) With Concurrent Accelerated Hyperfractionation Radiation Followed by Maintenance Therapy With OSI-774 for Stage III Non-Small Cell Lung Cancer
Brief Title: Erlotinib, Paclitaxel, and Carboplatin Combined With Radiation Therapy for Stage III Non-Small Cell Lung Cancer
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Nathan Pennell, MD, PhD (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor-Investigator, Nathan Pennell, MD, PhD, Principal Investigator, Case Comprehensive Cancer Center
Organization: Case Comprehensive Cancer Center (Other)
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: CCF5876; P30CA043703 (NIH); CCF-5876 (Other: Cleveland Clinic IRB)
Record Dates: First submitted 2006-01-16; First posted 2006-01-18 (Estimated); Results first posted 2020-07-20 (Actual); Last update posted 2020-07-20 (Actual); Status verified 2020-07

CONDITIONS: Lung Cancer
Keywords: stage IIIA non-small cell lung cancer; stage IIIB non-small cell lung cancer
MeSH Terms: conditions — Lung Neoplasms; Carcinoma, Non-Small-Cell Lung | interventions — Carboplatin; Erlotinib Hydrochloride; Paclitaxel; Radiotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Dose Level A (Experimental): Erlotinib, Paclitaxel, and Carboplatin with Radiation
  Dose Level A: 50 mg OSI-774/50 mg/m2 Paclitaxel/2 AUC Carboplatin
  Interventions: Drug: carboplatin; Drug: Erlotinib; Drug: paclitaxel; Procedure: conventional surgery; Radiation: radiation therapy
- Dose Level B (Experimental): Erlotinib, Paclitaxel, and Carboplatin with Radiation
  Dose Level B: 100 mg OSI-774/50 mg/m2 Paclitaxel/2 AUC Carboplatin
  Interventions: Drug: carboplatin; Drug: Erlotinib; Drug: paclitaxel; Procedure: conventional surgery; Radiation: radiation therapy
- Dose Level C (Experimental): Erlotinib, Paclitaxel, and Carboplatin with Radiation
  Dose Level C: 150 mg OSI-774/50 mg/m2 Paclitaxel/2 AUC Carboplatin
  Interventions: Drug: carboplatin; Drug: Erlotinib; Drug: paclitaxel; Procedure: conventional surgery; Radiation: radiation therapy

INTERVENTIONS:
Drug: carboplatin — AUC2 weekly x 3 weeks
  Other Names: Carbo
Drug: Erlotinib — Daily
  Other Names: OSI-774; Tarceva
Drug: paclitaxel — 50mg/m2/weekly x 3 weeks
Procedure: conventional surgery — conventional surgery
Radiation: radiation therapy — 150 cGy bid

SUMMARY:
RATIONALE: Erlotinib may stop the growth of tumor cells by blocking some of the enzymes needed for cell growth. Drugs used in chemotherapy, such as paclitaxel and carboplatin, work in different ways to stop the growth of tumor cells, either by killing the cells or by stopping them from dividing. Radiation therapy uses high-energy x-rays to kill tumor cells. Giving erlotinib, paclitaxel, and carboplatin together with radiation therapy before surgery may make the tumor smaller and reduce the amount of normal tissue that needs to be removed. Giving these treatments after surgery may kill any tumor cells that remain after surgery.

PURPOSE: This phase I/II trial is studying the best dose of erlotinib and the side effects of erlotinib, paclitaxel, and carboplatin when given together with radiation therapy and to see how well they work in treating patients who are undergoing surgery for stage III non-small cell lung cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Assess the safety and feasibility of erlotinib hydrochloride, paclitaxel, and carboplatin in combination with accelerated hyperfractionated radiotherapy in patients with stage IIIA or IIIB non-small cell lung cancer.
* Determine the maximum tolerated dose and recommended phase II dose of erlotinib hydrochloride in these patients.
* Assess the safety and tolerability of long-term maintenance erlotinib hydrochloride after completion of adjuvant chemoradiotherapy in these patients.

Secondary

* Evaluate the clinical and pathological response rate in these patients after neoadjuvant erlotinib hydrochloride, paclitaxel, carboplatin, and radiotherapy.
* Assess the impact of erlotinib hydrochloride on disease-free survival, overall survival, locoregional control, and distant metastatic control in these patients.

OUTLINE: This is an open-label, phase I dose-escalation study of erlotinib hydrochloride followed by a non-randomized phase II study.

Cohorts of 3-6 patients receive escalating doses of erlotinib hydrochloride until the maximum tolerated dose (MTD) is determined. The MTD is defined as the dose preceding that at which 2 of 3 or 2 of 6 patients experience dose-limiting toxicity.

* Phase I:

  * Neoadjuvant chemoradiotherapy: Patients receive oral erlotinib hydrochloride once daily on days 1-28 and paclitaxel IV over 1 hour and carboplatin IV over 30 minutes on days 1, 8, and 15 in the absence of disease progression or unacceptable toxicity. Patients concurrently undergo radiotherapy twice daily on days 1-5 and 8-12. Patients with complete response, partial response, or stable disease proceed to surgery. Patients who develop a medical contraindication to surgery (i.e., medically unresectable) receive a second course of erlotinib hydrochloride, paclitaxel, carboplatin, and radiotherapy as above within 2 weeks after completion of neoadjuvant chemoradiotherapy.

Cohorts of 3-6 patients receive escalating doses of erlotinib hydrochloride until the maximum tolerated dose (MTD) is determined. The MTD is defined as the dose preceding that at which 2 of 3 or 2 of 6 patients experience dose-limiting toxicity.

* Surgery: Within 4 weeks after completion of neoadjuvant chemoradiotherapy, patients undergo surgical resection and then proceed to adjuvant chemoradiotherapy.
* Adjuvant chemoradiotherapy: Within 6-8 weeks after surgery, patients receive a second course of erlotinib hydrochloride, paclitaxel, carboplatin, and radiotherapy as in neoadjuvant chemoradiotherapy.
* Maintenance therapy: All patients receive oral erlotinib hydrochloride once daily for 2 years in the absence of disease progression or unacceptable toxicity.

  * Phase II: Patients receive treatment as in phase I with erlotinib hydrochloride at the MTD.

After completion of study treatment, patients are followed periodically.

PROJECTED ACCRUAL: A total of 42 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically or cytologically confirmed non-small cell lung cancer

  * Surgically determined stage IIIA or IIIB disease
  * Histology from an involved mediastinal or supraclavicular lymph nodes alone will be allowed if a separate distal primary lesion is clearly evident on radiographs

    * Histological or cytological proof of mediastinal nodal involvement by mediastinoscopy, Chamberlain procedure, thoracoscopy, thoracotomy, or CT-guided biopsy is required except for cases of paralysis of left true vocal cord with separate left lung primary distinct from enlarged nodes > 1 cm in the anterior-posterior window seen on the CT scan
* Patients with N3 or T4 status must be evaluated and deemed potentially resectable after induction chemotherapy and radiation therapy
* Measurable and evaluable disease
* No malignant pleural effusion except for effusion visible only on CT scan and deemed too small to tap
* No pericardial effusion
* No small or mixed small cell/non-small cell lung cancer
* No massive lesions requiring radiation to the entire lung
* No metastatic cancer to the lungs

PATIENT CHARACTERISTICS:

* ECOG performance status 0-1
* WBC ≥ 3,000/mm^3
* Platelet count > 100,000/mm^3
* Serum creatinine ≤ 2.0 mg/dL
* Alkaline phosphatase, AST, and ALT < 2 times upper limit of normal
* Albumin > 3.0 g/dL
* Serum bilirubin < 1.5 mg/dL
* Adequate pulmonary function
* No clinical evidence of another uncontrolled malignancy
* No requirement for urgent therapy for severe local symptoms such as post-obstructive pneumonia

PRIOR CONCURRENT THERAPY:

* No prior chemotherapy, radiation therapy, or immunotherapy for lung cancer
* No prior surgery to treat the cancer

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2005-10; Primary Completion 2011-02 (Actual); Study Completion 2011-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Nathan Pennell, MD, Study Chair — Cleveland Clinic Taussig Cancer Institute, Case Comprehensive Cancer Center
Locations (1):
- Cleveland Clinic Taussig Cancer Institute, Case Comprehensive Cancer Center, Cleveland, Ohio, United States

REFERENCES:
- See also: Clinical trial summary from the National Cancer Institute's PDQ® database — http://clinicaltrials.gov/ct2/show/NCT00278148?term=ccf5876&rank=1

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 9 participants completed the phase I portion of the study. 3 of those subjects continued onto the phase II portion of the study and are included within the 26 participants.
Groups:
- Dose Level A: Dose Level A: 50 mg OSI-774/50 mg/m2 Paclitaxel/2 AUC Carboplatin
- Dose Level B: Dose Level B: 100 mg OSI-774/50 mg/m2 Paclitaxel/2 AUC Carboplatin
- Dose Level C: Dose Level C: 150 mg OSI-774/50 mg/m2 Paclitaxel/2 AUC Carboplatin
Period: Phase I - Dose Escalation
Arm/Group | Dose Level A | Dose Level B | Dose Level C
Started | 4 | 2 | 3
Completed | 4 | 2 | 3
Not Completed | 0 | 0 | 0
Period: Phase II - Expansion Phase
Arm/Group | Dose Level A | Dose Level B | Dose Level C
Started | 0 | 0 | 26 (Includes the 3 participants from phase I)
Completed | 0 | 0 | 20
Not Completed | 0 | 0 | 6
Not completed — Disease progression | 0 | 0 | 4
Not completed — Adverse Event | 0 | 0 | 2

BASELINE CHARACTERISTICS:
Groups:
- Erlotinib, Paclitaxel, and Carboplatin With Radiation: All participants that went on study at the three dose levels.
  Dose Level A: 50 mg OSI-774/50 mg/m2 Paclitaxel/2 AUC Carboplatin Dose Level B: 100 mg OSI-774/50 mg/m2 Paclitaxel/2 AUC Carboplatin Dose Level C: 150 mg OSI-774/50 mg/m2 Paclitaxel/2 AUC Carboplatin
Arm/Group | Erlotinib, Paclitaxel, and Carboplatin With Radiation
Number analyzed (Participants) | 32
Age, Continuous [Mean (Standard Deviation); unit: years] | 61 (10.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 18
  Male | 14
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 32
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 32
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 32

OUTCOME MEASURES:

1. Primary Outcome: Maximum Tolerated Dose of Erlotinib Hydrochloride (Phase I)
Description: The Phase I portion of this study is to determine the Maximum Tolerated Dose (MTD) of combining OSI-774 with the paclitaxel-carboplatin chemoradiation protocol and to assess the safety and feasiblity of this combination.
Time Frame: 2 weeks after surgery
Population: participants enrolled in the phase I portion of the study
Measure: Number; unit: mg daily
Groups:
- Erlotinib, Paclitaxel, and Carboplatin With Radiation: carboplatin: AUC2 weekly x 3 weeks
  Tarceva: Daily
  paclitaxel: 50mg/m2/weekly x 3 weeks
  conventional surgery: conventional surgery
  radiation therapy: 150 cGy bid
Arm/Group | Erlotinib, Paclitaxel, and Carboplatin With Radiation
Number analyzed (Participants) | 9
mg daily | 150

2. Primary Outcome: Tolerability of Long-term OSI-774 (Phase II)
Description: Number of patients who experienced grade >/= 3 toxicities on maintanance erolotinib (OSI-774)
Time Frame: 2 years
Population: Participants that completed adjuvant chemoradiation and maintenance erolotinib.
Measure: Count of Participants; unit: Participants
Arm/Group | Erlotinib, Paclitaxel, and Carboplatin With Radiation
Number analyzed (Participants) | 20
Participants
  grade 3 | 4
  less than grade 3 | 16

3. Secondary Outcome: Pathological Complete Response Rate
Description: Number of participants with an pathological complete response rate using the RECIST criteria.
  Complete response: Disappearance of all measurable and evaluable disease Partial response: A 30% or greater decline in the sum of the longest diameter of target lesions compared to the baseline measurement.
  Progressive disease: A 20% or greater increase in the sum of the longest diameter of the target lesions compared to the baseline.
  Stable disease: Disease that did not meet the criteria for a CR / PR or progressive disease.
Time Frame: 2 years
Population: Participants that participated in phase II portion of the study
Measure: Number; unit: participants
Arm/Group | Erlotinib, Paclitaxel, and Carboplatin With Radiation
Number analyzed (Participants) | 26
participants | 6

4. Secondary Outcome: Overall Survival
Description: Percent of participants still alive from the date of study entry to the date of the corresponding event (recurrence of death) or the date of final follow-up.
Time Frame: 3 years
Population: Participants that participated in the phase II of the study
Measure: Number; unit: percentage of participants
Arm/Group | Erlotinib, Paclitaxel, and Carboplatin With Radiation
Number analyzed (Participants) | 26
percentage of participants | 69

5. Secondary Outcome: Progression Free Survival (PFS)
Description: Months from the date of study entry to the date of the corresponding event (recurrence of death) or the date of final follow-up
Time Frame: 3 years
Population: Participants that participated in the phase II of the study
Measure: Median (Inter-Quartile Range); unit: months
Arm/Group | Erlotinib, Paclitaxel, and Carboplatin With Radiation
Number analyzed (Participants) | 26
months | 41.8 [9.2 to 51.8]

6. Secondary Outcome: Locoregional Control
Description: Estimated by the Kaplan-Meier method and summarized at various follow-up points as the number of patients remaining at risk, the event estimate, standard error, and median.From the date of study entry to the date of the corresponding event (recurrence of death) or the date of final follow-up, assessed up to 2 years
Time Frame: 2 years
Population: Data not collected
Groups:
- Erlotinib, Paclitaxel, and Carboplatin With Radiation: Participants received weekly Paclitaxel and Carboplatin (AUC 2) with daily oral Erlotinib for 28 days concurrent with twice daily thoracic radiation.
Arm/Group | Erlotinib, Paclitaxel, and Carboplatin With Radiation
Number analyzed (Participants) | 0

7. Secondary Outcome: Distant Control
Description: as for outcome 6
Time Frame: 2 years
Population: Data not collected
Arm/Group | Erlotinib, Paclitaxel, and Carboplatin With Radiation
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: Adverse events were collected over the duration of the study up to 3 years
Groups:
- Dose Level A:50 mg OSI-774/50 mg/m2: 50 mg OSI-774/50 mg/m2 Paclitaxel/2 AUC Carboplatin
- Dose Level B: 100 mg OSI-774/50 mg/m2: 100 mg OSI-774/50 mg/m2 Paclitaxel/2 AUC Carboplatin
- Dose Level C: 150 mg OSI-774/50 mg/m2: 150 mg OSI-774/50 mg/m2 Paclitaxel/2 AUC Carboplatin
Arm/Group | Dose Level A:50 mg OSI-774/50 mg/m2 | Dose Level B: 100 mg OSI-774/50 mg/m2 | Dose Level C: 150 mg OSI-774/50 mg/m2
All-Cause Mortality (participants affected / at risk) | 3/4 | 2/2 | 15/26
Serious Adverse Events (participants affected / at risk) | 2/4 | 1/2 | 9/26
Other Adverse Events (participants affected / at risk) | 4/4 | 2/2 | 26/26
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Dose Level A:50 mg OSI-774/50 mg/m2 (N=4) | Dose Level B: 100 mg OSI-774/50 mg/m2 (N=2) | Dose Level C: 150 mg OSI-774/50 mg/m2 (N=26)
Cardiac Arrhythmia (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Confusion (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (2)
Vomiting (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (2)
Memory impairment (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Vision-blurred vision (Eye disorders) | 1 (1) | 0 (0) | 0 (0)
Dyspnea (shortness of breath) (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (2)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Amylase (Investigations) | 0 (0) | 0 (0) | 1 (1)
Lipase (Investigations) | 0 (0) | 0 (0) | 1 (1)
Pain - Abdomen NOS (General disorders) | 0 (0) | 0 (0) | 1 (1)
Seizure (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Cholecystitis (Hepatobiliary disorders) | 0 (0) | 0 (0) | 1 (1)
Infection with unknown ANC - Skin (cellulitis) (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Hemorrhage, pulmonary/upper respiratory - Lung (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Thrombosis/thrombus/embolism (Vascular disorders) | 0 (0) | 1 (1) | 2 (3)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 2 (4)
Pneumonitis/pulmonary infiltrates (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Febrile neutropenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Dose Level A:50 mg OSI-774/50 mg/m2 (N=4) | Dose Level B: 100 mg OSI-774/50 mg/m2 (N=2) | Dose Level C: 150 mg OSI-774/50 mg/m2 (N=26)
Allergic reaction/hypersensitivity (including drug fever) (Immune system disorders) | 0 (0) | 1 (2) | 10 (15)
Allergic rhinitis (including sneezing, nasal stuffiness, postnasal drip) (Immune system disorders) | 0 (0) | 0 (0) | 6 (6)
Hemoglobin (Blood and lymphatic system disorders) | 2 (8) | 1 (5) | 20 (64)
Leukocytes (total WBC) (Blood and lymphatic system disorders) | 3 (6) | 1 (2) | 21 (57)
Lymphopenia (Blood and lymphatic system disorders) | 4 (16) | 2 (15) | 26 (142)
Neutrophils/granulocytes (ANC/AGC) (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 7 (12)
Platelets (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 9 (12)
Supraventricular and nodal arrhythmia - Atrial fibrillation (Cardiac disorders) | 0 (0) | 1 (1) | 4 (4)
Supraventricular and nodal arrhythmia - Sinus tachycardia (Cardiac disorders) | 0 (0) | 0 (0) | 2 (2)
Ventricular arrhythmia - Ventricular tachycardia (Cardiac disorders) | 0 (0) | 0 (0) | 2 (2)
Hypertension (Vascular disorders) | 0 (0) | 0 (0) | 2 (3)
Hypotension (Vascular disorders) | 0 (0) | 0 (0) | 3 (4)
Fatigue (asthenia, lethargy, malaise) (General disorders) | 4 (17) | 2 (10) | 21 (51)
Fever (in the absence of neutropenia, where neutropenia is defined as ANC <1.0 x 10e9/L) (General disorders) | 0 (0) | 0 (0) | 3 (3)
Insomnia (General disorders) | 0 (0) | 0 (0) | 7 (11)
Rigors/chills (General disorders) | 1 (1) | 0 (0) | 6 (10)
Sweating (diaphoresis) (General disorders) | 0 (0) | 0 (0) | 3 (3)
Weight loss (Investigations) | 1 (1) | 0 (0) | 10 (17)
Bruising (in absence of Grade 3 or 4 thrombocytopenia) (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 3 (4)
Cheilitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 3 (3)
Dry skin (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 10 (18)
Flushing (Vascular disorders) | 0 (0) | 0 (0) | 3 (5)
Hair loss/alopecia (scalp or body) (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 10 (11)
Nail changes (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 4 (6)
Rash/desquamation (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (3) | 13 (56)
Rash: acne/acneiform (Skin and subcutaneous tissue disorders) | 3 (7) | 2 (10) | 17 (65)
Rash: dermatitis associated with radiation - Chemoradiation (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 3 (3)
Anorexia (Metabolism and nutrition disorders) | 3 (6) | 1 (2) | 18 (28)
Constipation (Gastrointestinal disorders) | 2 (3) | 1 (1) | 11 (14)
Dehydration (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 5 (6)
Diarrhea (Gastrointestinal disorders) | 3 (6) | 2 (8) | 23 (79)
Distension/bloating, abdominal (Gastrointestinal disorders) | 0 (0) | 0 (0) | 4 (5)
Dysphagia (difficulty swallowing) (Gastrointestinal disorders) | 2 (5) | 2 (3) | 14 (20)
Esophagitis (Gastrointestinal disorders) | 3 (6) | 1 (2) | 6 (6)
Flatulence (Gastrointestinal disorders) | 0 (0) | 0 (0) | 3 (6)
Gastritis (including bile reflux gastritis) (Gastrointestinal disorders) | 0 (0) | 0 (0) | 2 (2)
Heartburn/dyspepsia (Gastrointestinal disorders) | 2 (2) | 0 (0) | 8 (13)
Mucositis/stomatitis (clinical exam) - Esophagus (Gastrointestinal disorders) | 1 (1) | 0 (0) | 4 (8)
Mucositis/stomatitis (clinical exam) - Oral cavity (Gastrointestinal disorders) | 1 (1) | 0 (0) | 12 (20)
Nausea (Gastrointestinal disorders) | 3 (6) | 2 (2) | 6 (13)
Taste alteration (dysgeusia) (Nervous system disorders) | 1 (1) | 0 (0) | 9 (17)
Vomiting (Gastrointestinal disorders) | 2 (2) | 0 (0) | 6 (19)
Hemorrhage, GI - Rectum (Gastrointestinal disorders) | 0 (0) | 0 (0) | 2 (2)
Hemorrhage, pulmonary/upper respiratory - Nose (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 8 (8)
Infection with normal ANC or Grade 1 or 2 neutrophils - Urinary tract NOS (Infections and infestations) | 0 (0) | 0 (0) | 2 (2)
Infection with unknown ANC - Pharynx (Infections and infestations) | 1 (1) | 0 (0) | 1 (1)
Opportunistic infection associated with >=Grade 2 Lymphopenia (Infections and infestations) | 0 (0) | 0 (0) | 2 (2)
Edema: limb (General disorders) | 0 (0) | 1 (1) | 1 (1)
Albumin, serum-low (hypoalbuminemia) (Metabolism and nutrition disorders) | 1 (1) | 1 (2) | 11 (19)
Alkaline phosphatase (Investigations) | 0 (0) | 1 (1) | 4 (4)
ALT, SGPT (serum glutamic pyruvic transaminase) (Blood and lymphatic system disorders) | 0 (0) | 1 (2) | 14 (18)
AST, SGOT(serum glutamic oxaloacetic transaminase) (Investigations) | 0 (0) | 1 (1) | 13 (20)
Bilirubin (hyperbilirubinemia) (Investigations) | 0 (0) | 0 (0) | 3 (4)
Calcium, serum-high (hypercalcemia) (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 4 (5)
Calcium, serum-low (hypocalcemia) (Metabolism and nutrition disorders) | 1 (1) | 1 (1) | 15 (33)
Creatinine (Investigations) | 0 (0) | 0 (0) | 2 (10)
Glucose, serum-high (hyperglycemia) (Metabolism and nutrition disorders) | 4 (15) | 2 (9) | 25 (136)
Glucose, serum-low (hypoglycemia) (Metabolism and nutrition disorders) | 0 (0) | 1 (2) | 2 (2)
Hemoglobinuria (Renal and urinary disorders) | 2 (2) | 1 (1) | 6 (12)
Phosphate, serum-low (hypophosphatemia) (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 5 (6)
Potassium, serum-high (hyperkalemia) (Metabolism and nutrition disorders) | 2 (2) | 1 (1) | 9 (10)
Potassium, serum-low (hypokalemia) (Metabolism and nutrition disorders) | 1 (1) | 1 (1) | 10 (13)
Sodium, serum-low (hyponatremia) (Metabolism and nutrition disorders) | 2 (6) | 1 (1) | 10 (17)
Uric acid, serum-high (hyperuricemia) (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 2 (3)
Muscle weakness, generalized or specific area (not due to neuropathy) - Extremity-lower (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 2 (2)
Muscle weakness, generalized or specific area (not due to neuropathy) - Whole body/generalized (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 2 (2)
Dizziness (Nervous system disorders) | 0 (0) | 1 (1) | 6 (12)
Mood alteration - Anxiety/Agitation (Psychiatric disorders) | 1 (1) | 0 (0) | 9 (13)
Mood alteration - Depression (Psychiatric disorders) | 0 (0) | 0 (0) | 3 (6)
mild paresthesias in hands/feet (Nervous system disorders) | 1 (1) | 1 (1) | 1 (2) — mild paresthesias in hands/feet
Neuropathy: motor (Nervous system disorders) | 0 (0) | 0 (0) | 2 (2)
Neuropathy: sensory (Nervous system disorders) | 1 (1) | 0 (0) | 6 (9) — tingling/burning of the fingers and toes
Dry eye syndrome (Eye disorders) | 0 (0) | 0 (0) | 2 (2)
Ocular surface disease (Eye disorders) | 0 (0) | 0 (0) | 2 (3)
Watery eye (epiphora, tearing) (Eye disorders) | 0 (0) | 0 (0) | 2 (3)
Pain - Back (Musculoskeletal and connective tissue disorders) | 2 (3) | 1 (2) | 3 (3)
Pain - Chest wall (Musculoskeletal and connective tissue disorders) | 2 (3) | 2 (3) | 5 (9)
Pain - Chest/thorax NOS (General disorders) | 1 (1) | 1 (2) | 4 (13)
Pain - Head/headache (Nervous system disorders) | 1 (1) | 0 (0) | 3 (3)
Pain - Joint (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 3 (4)
Pain - Muscle (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 3 (4)
Pain - Other NOS (General disorders) | 0 (0) | 0 (0) | 9 (30)
Pain - Skin (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 2 (2)
Pain - Throat/pharynx/larynx (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 2 (2)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (2) | 16 (28)
Dyspnea (shortness of breath) (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 1 (3) | 17 (27)
Hiccoughs (hiccups, singultus) (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 2 (3)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (2) | 1 (1)
Nasal cavity/paranasal sinus reactions (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 4 (8)
Voice changes/dysarthria (e.g., hoarseness, loss or alteration in voice, laryngitis) (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 8 (8)
Urinary frequency/urgency (Renal and urinary disorders) | 0 (0) | 0 (0) | 2 (2)
Phlebitis (including superficial thrombosis) (Vascular disorders) | 0 (0) | 0 (0) | 2 (2)
Thrombosis/thrombus/embolism (Vascular disorders) | 0 (0) | 1 (1) | 3 (4)

LIMITATIONS AND CAVEATS:
Some results were not assessible due to data not being collected.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No